CLINICAL TRIAL: NCT03074240
Title: A Prospective and Randomized Comparison of Ultrasound-guided Transversus Abdominis Plane Versus Rectus Sheath Blocks as a Primary Anesthetic for Abdominal Wall Surgery in Adults.
Brief Title: Abdominal Wall Block Study
Acronym: TAPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201602387 - V; OCR18951 (Other: University of Florida)
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Umbilical Hernia; Obesity
Keywords: Truncal block; Surgical anesthesia; Postoperative pain control
MeSH Terms: conditions — Hernia, Umbilical; Obesity | interventions — Anesthetics, General

STUDY DESIGN:
Intervention Model Description: Sixty subjects with be randomized to the TAPB or RSB arm upon enrollment, using randomized permutated blocks of six.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAPB Group (Active Comparator): Compare the instance in the TAPB group of intraoperative local anesthetic supplementation, analgesic administration, or conversion to general anesthesia when undergoing TAPB to anesthetize the abdominal wall.
  Interventions: Procedure: TAPB Group; Procedure: conversion to general anesthesia
- RSB Group (Active Comparator): Compare the instance in the RSB group of intraoperative local anesthetic supplementation, analgesic administration, or conversion to general anesthesia when undergoing RSB to anesthetize the abdominal wall.
  Interventions: Procedure: RSB Group; Procedure: conversion to general anesthesia

INTERVENTIONS:
Procedure: TAPB Group — Subjects allocated to the TAPB group will be monitored for instances of intraoperative local anesthetic supplementation, analgesic administration, or conversion to general anesthesia will be compared.
  Other Names: truncal peripheral nerve blocks; anesthetize the abdominal wall; ultrasound-guided regional anesthesia; Transversus abdominis plane blocks
  Arms: TAPB Group
Procedure: RSB Group — Subjects allocated to the RSB group will be monitored for instances of intraoperative local anesthetic supplementation, analgesic administration, or conversion to general anesthesia will be compared.
  Other Names: truncal peripheral nerve blocks; anesthetize the abdominal wall; ultrasound-guided regional anesthesia; rectus sheath blocks
  Arms: RSB Group
Procedure: conversion to general anesthesia — For those who do not respond to TAPB or RSB to allow for completion of the intended procedure.
  Other Names: general anesthetic

SUMMARY:
Compare the ability of the transversus abdominis plane block (TAPB) and rectus sheath block (RSB) to provide surgical anesthesia for overweight and obese patients undergoing umbilical hernia surgery.

DETAILED DESCRIPTION:
The purpose of this research study is to compare the ability of the TAPB and RSB to provide anesthesia for overweight and obese patients undergoing abdominal wall surgery. At the present time, this procedure is performed under general anesthesia, which often poses increased risks for overweight and obese individuals. It is not known if these blocks could be used to avoid the use of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age undergoing umbilical hernia repair
* Overweight and obese individuals (defined as a body mass index of ≥ 25 and 30 kg/m2, respectively)
* Ability to understand and provide informed consent

Exclusion Criteria:

* Patient refusal or inability to provide informed consent
* True allergy, not sensitivity, local anesthetics
* True allergy, not sensitivity, Propofol
* True allergy, not sensitivity, general anesthetic agents
* Pregnancy
* Severe hepatic impairment
* Evidence of infection at or near the proposed needle insertion site
* Any sensorimotor deficit, whether acute or chronic, as determined by the PI
* Chronic use of opioid medication

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Changes between the two groups to provide surgical anesthesia | Changes from baseline (pre-op) to 1 hour post-operative
  Assessed by the ability of the TAPB and RSB to provide primary surgical anesthesia

SECONDARY OUTCOMES:
Changes between the two groups assessed by post-operative pain control | Changes from baseline (post-operative) to 48 hours post-operative
  Assessed by instances of numerical rating scale pain scores (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: José R Soberón, MD, Principal Investigator — Malcom Randall VA Medical Center
Locations (1):
- Malcom Randall VA Medical Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No